CLINICAL TRIAL: NCT02282189
Title: Longitudinal Study of Oscillatory Positive Expiratory Pressure (oPEP) in Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROB0036
Record Dates: First submitted 2014-10-24; First posted 2014-11-04 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Sputum; Airway clearance therapy; Oscillatory Positive Expiratory Pressure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Off/on for 4 weeks followed by on/off for 4 weeks (Other): Subjects are randomized to either Oscillating Positive Expiratory Pressure device or no device for four weeks, then crossover for the following four weeks.
  Interventions: Device: Oscillating Positive Expiratory Pressure (Aerobika ®)

INTERVENTIONS:
Device: Oscillating Positive Expiratory Pressure (Aerobika ®) — The oPEP system combines positive expiratory pressure therapy and airway vibrations to help mobilize pulmonary secretions. oPEP therapy enforces a resistance to exhalation at the mouth, while the airway vibration technology transmits movements upstream during exhalation so that airway walls may become free from mucous. Subjects will take home the device and use four times daily during the active part of the study.
  Other Names: oPEP

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of four times daily oscillatory Positive Expiratory Pressure (oPEP) (Aerobika ®) use over 4 weeks in individuals with stable chronic obstructive pulmonary disease (COPD). The investigators hypothesize that daily oPEP use will significantly improve St. George's Respiratory Questionnaire (SGRQ) score, six-minute walk distance (6MWD) and forced expiratory volume in one second (FEV1) after four weeks of four times daily administration.

DETAILED DESCRIPTION:
Cough and sputum production is common in chronic obstructive pulmonary disease (COPD), both of which are associated with significant morbidity and other adverse clinical outcomes. Airway clearance techniques (ACTs) such as afforded by oscillatory Positive Expiratory Pressure (oPEP) (Aerobika ®) aim to remove sputum from the lungs, however evidence of their efficacy during stable disease is unclear.

The objective of this study is to evaluate the safety and efficacy of four times daily oPEP use over 4 weeks in individuals with stable COPD. The oPEP device combines positive expiratory pressure therapy and airway vibrations to help mobilize pulmonary secretions. oPEP therapy enforces a resistance to exhalation at the mouth while the airway vibration technology transmits movements upstream during exhalation so that airway walls may become free from mucus. An adjustable dial allows users to adjust the frequency and the flow resistance based on their individual needs. Subjects will take a device home and use four times daily during the active part of the study. We hypothesize that daily (Aerobika ®) use will significantly improve St. George's Respiratory Questionnaire (SGRQ) score, six-minute walk distance (6MWD) and forced expiratory volume in one second (FEV1) after four weeks of four times daily administration.

This is a randomized cross-over unblinded study in 15 subjects with COPD. All subjects will cross-over at four weeks of oPEP therapy or four weeks of no therapy. Each subject will visit the centre on five occasions (baseline, 2 weeks, 4 weeks (cross-over), 6 weeks and 8 weeks) for one hour each and will perform: 1) spirometry and plethysmography, 2) six-minute walk test (6MWT), and 3) health status evaluation using a self-administered St. George's Respiratory Questionnaire (SGRQ). Subjects will first provide written informed consent and will complete: 1) SGRQ after inhaling 2-4 puffs (200-400µg) of the short-acting bronchodilator (eg. Salbutamol), 2) plethysmography and spirometry 35±5 minutes post-salbutamol. Vital signs will be documented and subjects will rest for approximately 15 minutes before completing the six-minute walk test (6MWT) post-salbutamol. Subjects will be given an oPEP therapy system (Aerobika ®) to use at home, four times per day. Instruction and training on the use of the device will be given at the baseline visit. Subjects will be required to return the device upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 40-85 with a clinical diagnosis of chronic obstructive pulmonary disease (COPD)
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject is ambulatory and can perform the 6MWT
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater).
* FEV1 >25% predicted
* FVC > 25% predicted and >0.5L

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material. Capacity to consent will be determined by either Dr. McCormack at the time of the clinic visit or Sandra Blamires, the study coordinator.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Sputum Production | Weekly for eight weeks
  Change in sputum production from subject self-reported questionnaires performed weekly

SECONDARY OUTCOMES:
Six Minute Walk Distance (6MWD) | Baseline, 2-weeks, 4-weeks (cross-over), 6-weeks, 8-weeks
Pulmonary function measurements | Baseline, 2-weeks, 4-weeks (cross-over), 6-weeks, 8-weeks
  Pulmonary function measurements include FEV1 (Forced expiratory volume in 1 second); FVC (forced vital capacity); FEV1/FVC ratio; TLC (total lung capacity); RV (residual volume); DLCO (Diffusing capacity of the lung)
St. George's Respiratory Questionnaire (SGRQ) | Baseline, 2-weeks, 4-weeks (cross-over), 6-weeks, 8-weeks
Dyspnea (Patient Evaluation Questionnaire) | Completed weekly for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario; David G McCormack, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- Robarts Research Insitute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Svenningsen S, Paulin GA, Sheikh K, Guo F, Hasany A, Kirby M, Rezai RE, McCormack DG, Parraga G. Oscillatory Positive Expiratory Pressure in Chronic Obstructive Pulmonary Disease. COPD. 2016;13(1):66-74. doi: 10.3109/15412555.2015.1043523. Epub 2015 Oct 2. PMID 26430763